CLINICAL TRIAL: NCT06274944
Title: Nasogastric/Orogastric Tube Placement Confirmation in Neonates Utilizing Self-contained pH Device, a Feasibility Study
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2023-31694
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Premature Birth
Keywords: prematurity; nasogastric; orogastric
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Infants: Infants admitted to the University of Minnesota Masonic Children's Hospital neonatal intensive care unit.
  Interventions: Device: nasogastric tube placement pH confirmation device

INTERVENTIONS:
Device: nasogastric tube placement pH confirmation device — Each participation will get the contents tested by the novel device and the standard of care procedure.

SUMMARY:
This study is looking at using a self-contained pH device that will assist in confirming placement of a nasogastric or orogastric tube placed in the stomach of hospitalized infants.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the NICU at the University of Minnesota Masonic Children's Hospital, Minneapolis, MN requiring placement of an NG/OG tube are eligible to enroll.

Exclusion Criteria:

* Participant deemed unsuitable for study by the treating provider. Participants who are on the following medications: proton-pump inhibitor (PPI's) or H2 blockers within one week prior to the device assessment.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the University of Minnesota Masonic Children's Hospital neonatal intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
PH reading comparison | baseline
  Comparing the accuracy of the novel NG/OG tube placement device pH reading to the standard pH testing method.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strutt, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States